CLINICAL TRIAL: NCT00034879
Title: An Expanded Access Clinical Program With ZD1839 (IRESSA®) for Patients With Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: Iressa Expanded Access Program (EAP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0050
Expanded Access: Available
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Carcinoma; Non-small-cell Lung; Metastases; Neoplasm
Keywords: Locally advanced and/or metastatic non-operable; non-small cell lung cancer (stage III or IV); patients who have failed standard therapy.
MeSH Terms: conditions — Carcinoma; Neoplasm Metastasis; Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ZD1839 (Gefitinib)
  Other Names: Iressa

SUMMARY:
A program for patients with non small cell lung cancer who may benefit from Iressa, but cannot enter another clinical trial due to them not being eligible, or for whom no trials are available.

ELIGIBILITY:
Inclusion Criteria

For inclusion in this trial, patients must fulfill all of the following criteria:

* previous documented histologically or cytologically confirmed non-small cell lung cancer;
* locally advanced and/or metastatic non-operable non-small cell lung cancer (stage III or IV)patients who have received at least one course of standard systemic chemotherapy or radiation therapy or are ineligible for chemotherapy or radiotherapy or are ineligible or not a candidate for enrollment on another ZD1839 trial or who, in the Investigator's opinion, are not medically suitable for chemotherapy.
* age 18 years or older;
* written informed consent to participate in the trial.

Exclusion Criteria

Any of the following will exclude a patient from entering the trial:

* receiving concurrent radiotherapy, chemotherapy, or other systemic anti-cancer medication or any other investigational agent. * Non-cytotoxic or hormonal therapies for the adjuvant treatment of cancer or for previously treated cancers may be allowed per AstraZeneca permission;
* patients eligible for or previously enrolled on a ZD1839 blinded clinical trial protocol. Patients eligible for or previously enrolled on an open-label or unblinded ZD1839 clinical trial may be considered for acceptance into the Expanded Access Program with AstraZeneca permission;
* having other active malignancies;
* incomplete healing from previous oncologic or other major surgery;
* evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the trial;
* pregnancy or breast feeding (women of child-bearing potential).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iressa Medical Science Director, MD, Study Director — AstraZeneca
Locations (626):
- United States (626):
  - Research Site, Alabaster, Alabama
  - Research Site, Anniston, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Gadsen, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Montgomery, Alabama
  - Research Site, Anchorage, Alaska
  - Research Site, Fairbanks, Alaska
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Sedona, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Yuma, Arizona
  - Research Site, Bentonville, Arkansas
  - Research Site, Camden, Arkansas
  - Research Site, Fort Smith, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Arcadia, California
  - Research Site, Bakersfield, California
  - Research Site, Baldwin Park, California
  - Research Site, Bellflower, California
  - Research Site, Berkeley, California
  - Research Site, Burbank, California
  - Research Site, Campbell, California
  - Research Site, Chico, California
  - Research Site, Chino, California
  - Research Site, Chule Vista, California
  - Research Site, Concord, California
  - Research Site, Duarte, California
  - Research Site, Eureka, California
  - Research Site, Fairfield, California
  - Research Site, Fontana, California
  - Research Site, Fountain Valley, California
  - Research Site, Fresno, California
  - Research Site, Fullerton, California
  - Research Site, Gilroy, California
  - Research Site, Grass Valley, California
  - Research Site, Greenbrae, California
  - Research Site, La Jolla, California
  - Research Site, Lakewood, California
  - Research Site, LaVerne, California
  - Research Site, Loma Linda, California
  - Research Site, Long Beach, California
  - Research Site, Los Alamitos, California
  - Research Site, Los Angeles, California
  - Research Site, Los Gatos, California
  - Research Site, Marina Del Ray, California
  - Research Site, Mission Viejo, California
  - Research Site, Montebello, California
  - Research Site, Monterey, California
  - Research Site, Newport Beach, California
  - Research Site, Oakland, California
  - Research Site, Oceanside, California
  - Research Site, Orange, California
  - Research Site, Oxnard, California
  - Research Site, Palm Springs, California
  - Research Site, Palo Alto, California
  - Research Site, Panorama City, California
  - Research Site, Petaluma, California
  - Research Site, Pleasanton, California
  - Research Site, Rancho Mirage, California
  - Research Site, Redding, California
  - Research Site, Redondo Beach, California
  - Research Site, Redwood City, California
  - Research Site, Riverside, California
  - Research Site, Royal Grande, California
  - Research Site, Sacramento, California
  - Research Site, Salinas, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, San Jose, California
  - Research Site, San Luis Obispo, California
  - Research Site, San Mateo, California
  - Research Site, Santa Barbara, California
  - Research Site, Santa Clara, California
  - Research Site, Santa Cruz, California
  - Research Site, Santa Maria, California
  - Research Site, Santa Monica, California
  - Research Site, Simi Valley, California
  - Research Site, Soquel, California
  - Research Site, Stockton, California
  - Research Site, Sunnyvale, California
  - Research Site, Sylmar, California
  - Research Site, Tarzana, California
  - Research Site, Thousand Oaks, California
  - Research Site, Twentynine Palm, California
  - Research Site, Upland, California
  - Research Site, Vallejo, California
  - Research Site, Van Nuys, California
  - Research Site, Walnut Creek, California
  - Research Site, Westlake Village, California
  - Research Site, Woodland Hills, California
  - Research Site, Boulder, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Fort Collins, Colorado
  - Research Site, Longmont, Colorado
  - Research Site, Pueblo, Colorado
  - Research Site, Danbury, Connecticut
  - Research Site, Fairfield, Connecticut
  - Research Site, Greenwich, Connecticut
  - Research Site, Handen, Connecticut
  - Research Site, Hartford, Connecticut
  - Research Site, Manchester, Connecticut
  - Research Site, Middletown, Connecticut
  - Research Site, Milford, Connecticut
  - Research Site, New London, Connecticut
  - Research Site, New Milford, Connecticut
  - Research Site, Norwalk, Connecticut
  - Research Site, Norwich, Connecticut
  - Research Site, Stamford, Connecticut
  - Research Site, Torrington, Connecticut
  - Research Site, Trumbull, Connecticut
  - Research Site, Waterbury, Connecticut
  - Research Site, Lewes, Delaware
  - Research Site, Newark, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Boca Raton, Florida
  - Research Site, Boynton Beach, Florida
  - Research Site, Bradenton, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jupiter, Florida
  - Research Site, Key West, Florida
  - Research Site, Lake Worth, Florida
  - Research Site, Lakeland, Florida
  - Research Site, Leesburg, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Shores, Florida
  - Research Site, Naples, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Ocala, Florida
  - Research Site, Ocoee, Florida
  - Research Site, Orange Park, Florida
  - Research Site, Orlando, Florida
  - Research Site, Ormand Beach, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, Panama City, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Plantation, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Port Saint Lucie, Florida
  - Research Site, Saint Augustine, Florida
  - Research Site, Sanford, Florida
  - Research Site, Sarasota, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Stuart, Florida
  - Research Site, Tampa, Florida
  - Research Site, Tavares, Florida
  - Research Site, Vero Beach, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Albany, Georgia
  - Research Site, Athens, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Brunswick, Georgia
  - Research Site, Canton, Georgia
  - Research Site, Carrollton, Georgia
  - Research Site, Fort Gordon, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Roswell, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Thomasville, Georgia
  - Research Site, Tucker, Georgia
  - Research Site, Valdosta, Georgia
  - Research Site, Waycross, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Tripler AMC, Hawaii
  - Research Site, Wailuku, Hawaii
  - Research Site, Boise, Idaho
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, Idaho Falls, Idaho
  - Research Site, Arlington Heights, Illinois
  - Research Site, Aurora, Illinois
  - Research Site, Belleville, Illinois
  - Research Site, Berwyn, Illinois
  - Research Site, Champaign, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Chicago Heights, Illinois
  - Research Site, Danville, Illinois
  - Research Site, Decatur, Illinois
  - Research Site, Des Plaines, Illinois
  - Research Site, Elk Grove Village, Illinois
  - Research Site, Elmhurst, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Flossmore, Illinois
  - Research Site, Galesburg, Illinois
  - Research Site, Geneva, Illinois
  - Research Site, Harvey, Illinois
  - Research Site, Hinsdale, IL, Illinois
  - Research Site, Joliet, Illinois
  - Research Site, La Grange, Illinois
  - Research Site, Libertyville, Illinois
  - Research Site, Maywood, Illinois
  - Research Site, Moline, Illinois
  - Research Site, Naperville, Illinois
  - Research Site, Oak Lawn, Illinois
  - Research Site, Park Ridge, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, River Forest, Illinois
  - Research Site, Rockford, Illinois
  - Research Site, Skokie, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Urbana, Illinois
  - Research Site, Wheaton, Illinois
  - Research Site, Zion, Illinois
  - Research Site, Bloomington, Indiana
  - Research Site, Evansville, Indiana
  - Research Site, Fort Wayne, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Jasper, Indiana
  - Research Site, Merrillville, Indiana
  - Research Site, Michigan City, Indiana
  - Research Site, Muncie, Indiana
  - Research Site, Munster, Indiana
  - Research Site, New Albany, Indiana
  - Research Site, South Bend, Indiana
  - Research Site, Terre Haute, Indiana
  - Research Site, Ames, Iowa
  - Research Site, Bettendorf, Iowa
  - Research Site, Davenport, Iowa
  - Research Site, Des Moines, Iowa
  - Research Site, Iowa City, Iowa
  - Research Site, Mason City, Iowa
  - Research Site, Sioux City, Iowa
  - Research Site, Waterloo, Iowa
  - Research Site, Hays, Kansas
  - Research Site, Hutchinson, Kansas
  - Research Site, Kansas City, Kansas
  - Research Site, Lawrence, Kansas
  - Research Site, Lenexa, Kansas
  - Research Site, Topeka, Kansas
  - Research Site, Witchita, Kansas
  - Research Site, Ashland, Kentucky
  - Research Site, Danville, Kentucky
  - Research Site, Hazard, Kentucky
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Paducah, Kentucky
  - Research Site, Pikeville, Kentucky
  - Research Site, Trenton, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Debque, Louisiana
  - Research Site, Lafayette, Louisiana
  - Research Site, Lake Charles, Louisiana
  - Research Site, Metairie, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Slidell, Louisiana
  - Research Site, Thiodaux, Louisiana
  - Research Site, Bangor, Maine
  - Research Site, Scarborough, Maine
  - Research Site, Waterville, Maine
  - Research Site, York Village, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Cumberland, Maryland
  - Research Site, Olney, Maryland
  - Research Site, Rockville, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Waldorf, Maryland
  - Research Site, Beverly, Massachusetts
  - Research Site, Boston, Massachusetts
  - Research Site, Brockton, Massachusetts
  - Research Site, Burlington, Massachusetts
  - Research Site, Chicopee, Massachusetts
  - Research Site, Lowell, Massachusetts
  - Research Site, Mansfield, Massachusetts
  - Research Site, Medford, Massachusetts
  - Research Site, Pittsfield, Massachusetts
  - Research Site, Quincy, Massachusetts
  - Research Site, South Weymouth, Massachusetts
  - Research Site, Springfield, Massachusetts
  - Research Site, Stoneham, Massachusetts
  - Research Site, Taunton, Massachusetts
  - Research Site, Walpole, Massachusetts
  - Research Site, Wareham, Massachusetts
  - Research Site, Wellesley, Massachusetts
  - Research Site, Woburn, Massachusetts
  - Research Site, Worchester, Massachusetts
  - Research Site, Battle Kreek, Michigan
  - Research Site, Bay City, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Free Soil, Michigan
  - Research Site, Golfport, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Grosse Point Woods, Michigan
  - Research Site, Iron Mountain, Michigan
  - Research Site, Jackson, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Lapeer, Michigan
  - Research Site, Marquette, Michigan
  - Research Site, Midland, Michigan
  - Research Site, Mount Clemens, Michigan
  - Research Site, Muskegon, Michigan
  - Research Site, Petoskey, Michigan
  - Research Site, Poplar Buff, Michigan
  - Research Site, Port Huron, Michigan
  - Research Site, Roseville, Michigan
  - Research Site, Royal Oak, Michigan
  - Research Site, Saint Joseph, Michigan
  - Research Site, Southfield, Michigan
  - Research Site, Traverse City, Michigan
  - Research Site, Ypsilanti, Michigan
  - Research Site, Alexandria, Minnesota
  - Research Site, Bemidji, Minnesota
  - Research Site, Brainerd, Minnesota
  - Research Site, Duluth, Minnesota
  - Research Site, Maplewood, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Roseville, Minnesota
  - Research Site, Saint Cloud, Minnesota
  - Research Site, Saint Louis Park, Minnesota
  - Research Site, Hattiesburg, Mississippi
  - Research Site, Jackson, Mississippi
  - Research Site, Pascagoula, Mississippi
  - Research Site, Tupelo, Mississippi
  - Research Site, Branson, Missouri
  - Research Site, Chesterfield, Missouri
  - Research Site, Columbia, Missouri
  - Research Site, Creve Coeus, Missouri
  - Research Site, Joplin, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Poplar Bluff, Missouri
  - Research Site, Saint Charles, Missouri
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Billings, Montana
  - Research Site, Great Falls, Montana
  - Research Site, Helena, Montana
  - Research Site, Grand Island, Nebraska
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Hooksett, New Hampshire
  - Research Site, Lebanon, New Hampshire
  - Research Site, Nashua, New Hampshire
  - Research Site, Belleville, New Jersey
  - Research Site, Denville, New Jersey
  - Research Site, Elizabeth, New Jersey
  - Research Site, Englewood, New Jersey
  - Research Site, Flemington, New Jersey
  - Research Site, Galloway, New Jersey
  - Research Site, Hackensack, New Jersey
  - Research Site, Little Silver, New Jersey
  - Research Site, Livingston, New Jersey
  - Research Site, Long Branch, New Jersey
  - Research Site, Mahwah, New Jersey
  - Research Site, Manasquan, New Jersey
  - Research Site, Montclair, New Jersey
  - Research Site, Morristown, New Jersey
  - Research Site, Mount Holly, New Jersey
  - Research Site, New Brunswick, New Jersey
  - Research Site, Newark, New Jersey
  - Research Site, Old Bridge, New Jersey
  - Research Site, Paramus, New Jersey
  - Research Site, Phillipsburg, New Jersey
  - Research Site, Plainfield, New Jersey
  - Research Site, Pompton Plains, New Jersey
  - Research Site, Princeton, New Jersey
  - Research Site, Red Bank, New Jersey
  - Research Site, Somerset, New Jersey
  - Research Site, Summit, New Jersey
  - Research Site, Teaneck, New Jersey
  - Research Site, Union, New Jersey
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Westwood, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Farmington, New Mexico
  - Research Site, Las Cruces, New Mexico
  - Research Site, Roswell, New Mexico
  - Research Site, Santa Fe, New Mexico
  - Research Site, Albany, New York
  - Research Site, Bay Shore, New York
  - Research Site, Bayside, New York
  - Research Site, Bronxville, New York
  - Research Site, Brooklyn, New York
  - Research Site, Buffalo, New York
  - Research Site, Cooperstown, New York
  - Research Site, East Setauket, New York
  - Research Site, East Syracuse, New York
  - Research Site, Flushing, New York
  - Research Site, Fresh Meadows, New York
  - Research Site, Geneseo, New York
  - Research Site, Glen Cove, New York
  - Research Site, Glens Falls, New York
  - Research Site, Goshen, New York
  - Research Site, Great Neck, New York
  - Research Site, Harris, New York
  - Research Site, Huntington, New York
  - Research Site, Huntington Station, New York
  - Research Site, Johnson City, New York
  - Research Site, Lake Success, New York
  - Research Site, Malone, New York
  - Research Site, Merrick, New York
  - Research Site, Mineola, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New Rochelle, New York
  - Research Site, New York, New York
  - Research Site, Northport, New York
  - Research Site, Nyack, New York
  - Research Site, Pomona, New York
  - Research Site, Port Washington, New York
  - Research Site, Riverhead, New York
  - Research Site, Rochester, New York
  - Research Site, Rockville Centre, New York
  - Research Site, Schenectady, New York
  - Research Site, Staten Island, New York
  - Research Site, Suffern, New York
  - Research Site, Syosset, New York
  - Research Site, The Bronx, New York
  - Research Site, Utica, New York
  - Research Site, Valhalla, New York
  - Research Site, Valley Stream, New York
  - Research Site, West Islip, New York
  - Research Site, White Plains, New York
  - Research Site, Wiliamsville, New York
  - Research Site, Williamsville, New York
  - Research Site, Woodbury, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Boone, North Carolina
  - Research Site, Burlington, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Concord, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Elizabeth, North Carolina
  - Research Site, Fayetteville, North Carolina
  - Research Site, Forest City, North Carolina
  - Research Site, Goldsboro, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Kinston, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Valdese, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Bismarck, North Dakota
  - Research Site, Fargo, North Dakota
  - Research Site, Grand Forks, North Dakota
  - Research Site, Akron, Ohio
  - Research Site, Barberton, Ohio
  - Research Site, Bryan, Ohio
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Fairfield, Ohio
  - Research Site, Finley, Ohio
  - Research Site, Independence, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Mansfield, Ohio
  - Research Site, Mentor, Ohio
  - Research Site, Middleburg Heights, Ohio
  - Research Site, Middletown, Ohio
  - Research Site, Sandusky, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Troy, Ohio
  - Research Site, Warrensville Heights, Ohio
  - Research Site, Wooster, Ohio
  - Research Site, Youngstown, Ohio
  - Research Site, Zanesville, Ohio
  - Research Site, Enid, Oklahoma
  - Research Site, Lawton, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Ponca City, Oklahoma
  - Research Site, Stillwater, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Bend, Oregon
  - Research Site, Coos Bay, Oregon
  - Research Site, Corvallis, Oregon
  - Research Site, Eugene, Oregon
  - Research Site, Klamath, Oregon
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Salem, Oregon
  - Research Site, Tualatin, Oregon
  - Research Site, Allentown, Pennsylvania
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Bryn Mawr, Pennsylvania
  - Research Site, Butler, Pennsylvania
  - Research Site, Cellarsville, Pennsylvania
  - Research Site, Danville, Pennsylvania
  - Research Site, Drexel Hill, Pennsylvania
  - Research Site, Dunmore, Pennsylvania
  - Research Site, East Stroudsburg, Pennsylvania
  - Research Site, Easton, Pennsylvania
  - Research Site, Ephrata, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Franklin, Pennsylvania
  - Research Site, Greensburg, Pennsylvania
  - Research Site, Harrisburg, Pennsylvania
  - Research Site, Hazleton, Pennsylvania
  - Research Site, Kingston, Pennsylvania
  - Research Site, Kittanning, Pennsylvania
  - Research Site, Lancaster, Pennsylvania
  - Research Site, Langhorne, Pennsylvania
  - Research Site, Langhorn, Pennsylvania
  - Research Site, Lemoyne, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Phoenixville, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Pottstown, Pennsylvania
  - Research Site, Pottsville, Pennsylvania
  - Research Site, Saint Marys, Pennsylvania
  - Research Site, Sayre, Pennsylvania
  - Research Site, Scranton, Pennsylvania
  - Research Site, State College, Pennsylvania
  - Research Site, West Reading, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Pawtucket, Rhode Island
  - Research Site, Providence, Rhode Island
  - Research Site, Warwick, Rhode Island
  - Research Site, Westerly, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Florence, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Spartenburg, South Carolina
  - Research Site, Aberdeen, South Dakota
  - Research Site, Rapid City, South Dakota
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Chattanooga, Tennessee
  - Research Site, Collierville, Tennessee
  - Research Site, Jackson, Tennessee
  - Research Site, Johnson City, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Abilene, Texas
  - Research Site, Amarillo, Texas
  - Research Site, Arlington, Texas
  - Research Site, Austin, Texas
  - Research Site, Baytown, Texas
  - Research Site, Beaumont, Texas
  - Research Site, Bryan, Texas
  - Research Site, Corpus Christi, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Fredricksburg, Texas
  - Research Site, Garland, Texas
  - Research Site, Houston, Texas
  - Research Site, Irving, Texas
  - Research Site, Lewisville, Texas
  - Research Site, Lubbock, Texas
  - Research Site, McAllen, Texas
  - Research Site, Mesquite, Texas
  - Research Site, Midland, Texas
  - Research Site, New Braunfels, Texas
  - Research Site, Paris, Texas
  - Research Site, Pasadena, Texas
  - Research Site, Plano, Texas
  - Research Site, Richmond, Texas
  - Research Site, San Antonio, Texas
  - Research Site, San Marcos, Texas
  - Research Site, Sherman, Texas
  - Research Site, Temple, Texas
  - Research Site, Tyler, Texas
  - Research Site, Victoria, Texas
  - Research Site, Waco, Texas
  - Research Site, Walla Walla, Texas
  - Research Site, Webster, Texas
  - Research Site, Ivins, Utah
  - Research Site, Ogden, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Bennington, Vermont
  - Research Site, Rutland, Vermont
  - Research Site, Abington, Virginia
  - Research Site, Charlottesville, Virginia
  - Research Site, Chesapeake, Virginia
  - Research Site, Danville, Virginia
  - Research Site, Fairfax, Virginia
  - Research Site, Fredericksburg, Virginia
  - Research Site, Hampton, Virginia
  - Research Site, Lynchburg, Virginia
  - Research Site, Newport News, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Portsmouth, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Williamsburg, Virginia
  - Research Site, Woodridge, Virginia
  - Research Site, Auburn, Washington
  - Research Site, Bremerton, Washington
  - Research Site, Kennewick, Washington
  - Research Site, Kirkland, Washington
  - Research Site, Mount Vernon, Washington
  - Research Site, Olympia, Washington
  - Research Site, Renton, Washington
  - Research Site, Seattle, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Vancouver, Washington
  - Research Site, Clarksburg, West Virginia
  - Research Site, Huntington, West Virginia
  - Research Site, Morgantown, West Virginia
  - Research Site, Princeton, West Virginia
  - Research Site, Wheeling, West Virginia
  - Research Site, Appleton, Wisconsin
  - Research Site, Eau Claire, Wisconsin
  - Research Site, Green Bay, Wisconsin
  - Research Site, Janesville, Wisconsin
  - Research Site, La Crosse, Wisconsin
  - Research Site, Madison, Wisconsin
  - Research Site, Manitowoc, Wisconsin
  - Research Site, Marshfield, Wisconsin
  - Research Site, Milwaukee, Wisconsin
  - Research Site, Racine, Wisconsin
  - Research Site, Rhinelander, Wisconsin
  - Research Site, Sheboygan, Wisconsin
  - Research Site, Waukesha, Wisconsin
  - Research Site, Wausau, Wisconsin
  - Research Site, Cheyenne, Wyoming